CLINICAL TRIAL: NCT02548325
Title: Prevalence of Hepatitis B in Vallés Occidental. Observational Multicentric Study
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Mireia Miquel-Planas, phD, Corporacion Parc Tauli
Other Study IDs: CorporacionPT
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Not apply — None. Just registration epidemiology dates

SUMMARY:
The aim of this study is to evaluate the prevalence of hepatitis B in Vallés Occidental. Also, describe the stage of the disease, and whether if they are under medical treatment or not.

DETAILED DESCRIPTION:
The hepatitis B virus ( HBV ) is a global health problem . It is estimated that in the world there are about 350-400 million carriers of HBV surface antigen ( HBsAg ) 1 .

The prevalence in Spain is estimated at a 2-7 % and is considered a second intermediate prevalence.

For over 20 years, has carried out a program of primary prevention through universal vaccination against hepatitis B including it in the childhood vaccination schedule and has already been observed that in some estudi3 the prevalence has declined . For this reason , we want to evaluate what is the currently prevalence in our area of influence. There aren't recent studies to assess what is the current status of these patients ( how many , what risk factors which needs of treatment and with answer ...)

ELIGIBILITY:
Inclusion Criteria:

* Patients with HBsAg + visited in Digestive/Hepatology outpatient visits and Hepatology of the participating hospitals

Exclusion Criteria:

* Patients < 18 aged
* Duplicity on record

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The are Included consecutively for one year ( 1 June 2014 to 31 May 2015 ) all patients who are in the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
prevalence hepatitis B | 12 months

SECONDARY OUTCOMES:
stage of the disease and if they are in treatment or not | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Mútua de Terrassa, Terrassa, Barcelona, Spain